CLINICAL TRIAL: NCT04878731
Title: A PHASE 1, SINGLE-ARM, OPEN-LABEL, NON-RANDOMIZED, NON-CONTROLLED MULTICENTER STUDY TO EVALUATE THE PHARMACOKINETICS, PHARMACODYNAMICS, SAFETY, AND TOLERABILITY OF A SINGLE SUBCUTANEOUS DOSE OF PF-06741086 IN CHINESE ADULT PARTICIPANTS WITH SEVERE HEMOPHILIA
Brief Title: Study to Evaluate Safety and Tolerability of a Single Dose of PF-06741086 in Chinese Adult Participants With Severe Hemophilia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B7841010
Record Dates: First submitted 2021-04-16; First posted 2021-05-07 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2022-08

CONDITIONS: Severe Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — marstacimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): PF-06741086 300mg subcutaneous(SC)
  Interventions: Biological: PF-06741086

INTERVENTIONS:
Biological: PF-06741086 — single dose SC injection of 300 mg PF-06741086

SUMMARY:
This Phase 1 study will be a single-arm, open-label, non-randomized, non-controlled investigation of the safety, tolerability, pharmacokinetics, and pharmacodynamics of PF-06741086 in Chinese adult participants with severe hemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be male and 18 to <75 years of age with a minimum body weight of 30 kg at screening.
* Participants with a diagnosis of severe hemophilia A or B (FVIII or FIX activity <1%, respectively)
* Participants without inhibitor must also meet the following criteria:

  * No detectable or documented history of inhibitors
  * Participants with on-demand treatment regimen with ≥6 acute bleeding episodes (spontaneous or traumatic) that required coagulation factor infusion during the 4 months period prior to enrollment and willing to continue to receive on demand treatment during the study.
* Participants with Inhibitor must also meet the following criteria:

  * Documentation of current high titer inhibitor (≥5 BU/mL) or current low titer inhibitor (<5 BU/mL) refractory to FVIII or FIX replacement and with FVIII or FIX recovery <60% of expected within previous 4 months prior to screening.
  * Participants with on-demand treatment regimen with ≥6 bleeding episodes (spontaneous and/or traumatic) necessitating treatment with bypass factor for at least 4 months prior to screening and willing to continue to receive on-demand treatment during the study.

Exclusion Criteria:

* Previous or current treatment for and/or history of coronary artery diseases, venous or arterial thrombosis or ischemic disease
* Known planned surgical procedure during the planned study period.
* Known hemostatic defect other than hemophilia A or B.
* Abnormal renal or hepatic function
* Current unstable liver or biliary disease
* Abnormal hematologic parameters
* Abnormal coagulation activity
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator.
* Corrected QT interval (QTc) >450 msec for male participants or QTc >480 msec in participants with bundle branch block.
* Individuals with hypersensitivity or an allergic reaction to hamster protein or other components of the study intervention.
* A positive urine drug screen
* Current routine prophylaxis with bypassing agent or non coagulation factor-replacement therapy (eg, emicizumab)
* Regular, concomitant therapy with immunomodulatory drugs
* Ongoing or planned use of immune tolerance induction or prophylaxis with FVIII or FIX replacement during the study.
* Participation in other studies involving investigational drug(s) within 30 days (or as determined by local requirements) or 5 half-lives prior to study entry and/or during study participation.
* CD4 cell count ≤200/uL if human immunodeficiency virus (HIV)-positive
* Baseline ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are Pfizer employees, including their family members, directly involved in the conduct of the study

Ages: 18 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Institute of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7841010

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 6 participants were enrolled and received a single dose of marstacimab 300 mg.
Groups:
- PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose: Participants received a single SC injection of marstacimab 300 mg on Study Day 1.
Period: Overall Study
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants enrolled in the study who received the study intervention.
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 31.5 [27 to 34]
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0
  18-64 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 6
  Other (Not Chinese) | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0
  Black or African American | 0
  Asian | 6
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with study treatment. TEAEs=AEs that started during the effective duration of treatment regardless of whether a similar event existed at baseline. Grades of AEs were defined by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 5.0. Grade 1=asymptomatic/mild symptoms, clinical or diagnostic observations only, intervention not indicated;Grade 2=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activity of daily living (ADL);Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL;Grade 4=events with life-threatening consequences, urgent intervention indicated;Grade 5= death related to AE.Treatment-related TEAEs were determined by investigator.
Time Frame: Day 1 to Day 42
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Participants
  All-Causality TEAEs | 1
  Treatment-Related TEAEs | 0
  All-Causality Severe TEAEs | 0

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect. Treatment-related SAEs were determined by the investigator.
Time Frame: Day 1 to Day 42
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Participants | 0

3. Primary Outcome: Number of Participants With Maximum Grade 3 or 4 or 5 TEAEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with study treatment. TEAEs=AEs that started during the effective duration of treatment regardless of whether a similar event existed in the baseline period. Grades of AEs were defined by NCI CTCAE version 5.0. Grade 1=asymptomatic/mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activity of daily living (ADL); Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4=events with life-threatening consequences, urgent intervention indicated; Grade 5= death related to AE. Treatment-related TEAEs were determined by the investigator.
Time Frame: Day 1 to Day 42
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Participants | 0

4. Primary Outcome: Number of Participants With TEAEs Leading to Permanent or Temporary Discontinuation From Study
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with study treatment. TEAEs=AEs that started during the effective duration of treatment regardless of whether a similar event of equal or greater severity existed in the baseline period. Grades of AEs were defined by NCI CTCAE version 5.0. Grade 1=asymptomatic/mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activity of daily living (ADL); Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4=events with life-threatening consequences, urgent intervention indicated; Grade 5= death related to AE. Treatment-related TEAEs were determined by the investigator.
Time Frame: Day 1 to Day 42
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Participants | 0

5. Primary Outcome: Number of Participants With Laboratory Abnormalities Without Regard to Baseline Abnormality
Description: Laboratory assessments included chemistry, hematology, Prothrombin Time/International Normalized Ratio (PT/INR), Activated Partial Thromboplastin Time (APTT), urinalysis, fibrinogen, Antithrombin III (ATIII) activity, and Cardiac Troponin I (cTnI). Laboratory test abnormalities reported by at least 1 participant are reported in this outcome measure. ULN = upper limit of normal.
Time Frame: Day 1 to Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Participants
  APTT >1.1 x ULN | 6
  Urine hemoglobin >=1 | 1
  Urobilinogen >=1 | 2

6. Primary Outcome: Mean Absolute Value of Prothrombin Time (PT) / International Normalized Ratio (INR)
Description: PT is one of the laboratory tests to evaluate the ability of blood clotting. The INR is derived from PT which is calculated as a ratio of a participant's PT to a control PT standardized for the potency of the thromboplastin reagent developed by the World Health Organization (WHO) using the following formula: INR = Participant PT / Control PT. Blood samples were obtained to evaluate PT/INR.
Time Frame: Day 1, Day 2, Day 7, Day 14, Day 21, Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
ratio
  Day 1 | 1.000 (0.0790)
  Day 2 | 0.990 (0.0632)
  Day 7 | 0.972 (0.0549)
  Day 14 | 0.960 (0.0690)
  Day 21 | 0.982 (0.0902)
  Day 28 | 0.988 (0.0920)

7. Primary Outcome: Change From Baseline in PT/INR at Days 2, 7, 14, 21 and 28
Description: PT is one of the laboratory tests to evaluate the ability of blood clotting. The INR is derived from PT which is calculated as a ratio of a participant's PT to a control PT standardized for the potency of the thromboplastin reagent developed by the WHO using the following formula: INR = Participant PT / Control PT. Blood samples were obtained to evaluate PT/INR.
Time Frame: Baseline (Day 1), Day 2, Day 7, Day 14, Day 21, Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Ratio
  Day 2 | -0.010 (0.0363)
  Day 7 | -0.028 (0.0611)
  Day 14 | -0.040 (0.0379)
  Day 21 | -0.018 (0.0492)
  Day 28 | -0.012 (0.0741)

8. Primary Outcome: Mean Absolute Value of Activated Partial Thromboplastin Time (APTT)
Description: The APTT is a screening test that helps evaluate a person's ability to appropriately form blood clots. It measures the number of seconds it takes for a clot to form in a sample of blood after substances (reagents) are added. Blood samples were obtained to evaluate APTT.
Time Frame: Day 1, Day 2, Day 7, Day 14, Day 21, Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: second
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
second
  Day 1 | 85.38 (14.377)
  Day 2 | 87.15 (15.473)
  Day 7 | 87.78 (14.376)
  Day 14 | 80.95 (17.521)
  Day 21 | 64.10 (21.833)
  Day 28 | 68.92 (16.144)

9. Primary Outcome: Change From Baseline in APTT at Days 2, 7, 14, 21 and 28
Description: as for outcome 8
Time Frame: Baseline (Day 1), Day 2, Day 7, Day 14, Day 21, Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: Second
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Second
  Day 2 | 1.77 (6.431)
  Day 7 | 2.40 (7.294)
  Day 14 | -4.43 (16.987)
  Day 21 | -21.28 (16.632)
  Day 28 | -16.47 (13.733)

10. Primary Outcome: Mean Absolute Value of Fibrinogen
Description: Fibrinogen is a protein, specifically a clotting factor (factor I), that is essential for proper blood clot formation. Blood samples were obtained to evaluate the amount of fibrinogen.
Time Frame: Day 1, Day 2, Day 7, Day 14, Day 21, Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
milligram per deciliter (mg/dL)
  Day 1 | 284.3 (61.68)
  Day 2 | 267.0 (52.37)
  Day 7 | 249.5 (72.82)
  Day 14 | 284.0 (50.12)
  Day 21 | 267.7 (30.18)
  Day 28 | 273.2 (43.73)

11. Primary Outcome: Change From Baseline in Fibrinogen at Days 2, 7, 14, 21 and 28
Description: as for outcome 10
Time Frame: Baseline (Day 1), Day 2, Day 7, Day 14, Day 21, Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
mg/dL
  Day 2 | -17.3 (26.82)
  Day 7 | -34.8 (27.02)
  Day 14 | -0.3 (39.73)
  Day 21 | -16.7 (39.33)
  Day 28 | -11.2 (74.66)

12. Primary Outcome: Mean Absolute Value of Antithrombin III (ATIII)
Description: ATIII is a nonvitamin K-dependent protease that inhibits coagulation by lysing thrombin and factor Xa. The antithrombin activity test measures how well the protein inhibits thrombin, with a reference range of 75% - 125%. Blood samples were obtained to evaluate ATIII activity.
Time Frame: Day 1, Day 2, Day 7, Day 14, Day 21, Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: percent of antithrombin III activity
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
percent of antithrombin III activity
  Day 1 | 92.75 (6.498)
  Day 2 | 88.68 (3.939)
  Day 7 | 94.07 (4.384)
  Day 14 | 97.98 (6.386)
  Day 21 | 96.10 (3.949)
  Day 28 | 97.18 (7.885)

13. Primary Outcome: Change From Baseline in ATIII at Days 2, 7, 14, 21 and 28
Description: as for outcome 12
Time Frame: Baseline (Day 1), Day 2, Day 7, Day 14, Day 21, Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: percent of antithrombin III activity
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
percent of antithrombin III activity
  Day 2 | -4.07 (4.399)
  Day 7 | 1.32 (5.739)
  Day 14 | 5.23 (7.655)
  Day 21 | 3.35 (5.899)
  Day 28 | 4.43 (6.207)

14. Primary Outcome: Mean Absolute Value of Cardiac Troponin I (cTnI)
Description: cTnI is one of the cardiac regulatory proteins that control the calcium mediated interaction between actin and myosin, and is considered a specific marker for cardiac damage. Blood samples were obtained to evaluate the amount of cTnI.
Time Frame: Day 1, Day 2, Day 4
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention. Number of Participants Analyzed = Number of participants evaluable for this outcome measure. Number Analyzed = number of participants evaluable at the specific time point.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
nanogram per milliliter (ng/mL)
  Day 1 | 0.0250 (0.00000)
  Day 2: number analyzed (Participants) | 5
  Day 2 | 0.0250 (0.00000)
  Day 4 | 0.0250 (0.00000)

15. Primary Outcome: Change From Baseline in cTnI at Days 2 and 4
Description: as for outcome 14
Time Frame: Baseline (Day 1), Day 2, Day 4
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
ng/mL
  Day 2: number analyzed (Participants) | 5
  Day 2 | 0.0000 (0.0000)
  Day 4 | 0.0000 (0.00000)

16. Primary Outcome: Number of Participants With Vital Signs Data Meeting Categorical Criteria of Potential Clinical Concern
Description: Vital signs measurements included blood pressure (BP), pulse rate, respiratory rate and oral temperature. Categorical classes for vital signs of potential clinical concern included: (1) systolic BP - minimum (min) value <90 mmHg, maximum (max) decrease/increase from baseline >=30 mmHg; (2) diastolic BP - min value <50 mmHg, max decrease/increase from baseline >=20 mmHg; (3) supine pulse rate - min <40 beat per minute (bpm) or max >120 bpm; (4) standing pulse rate - min <40 bpm or max >140 bpm; (5) oral temperature > 38.5 celsius degree (°C). BPs were measured in a supine position so standing BPs were not evaluated and not reported.
Time Frame: Day 1 to Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Participants
  Supine systolic BP value <90 mmHg | 0
  Supine systolic BP increase from baseline >=30 mmHg | 0
  Supine systolic BP decrease from baseline >=30 mmHg | 0
  Supine diastolic BP value <50 mmHg | 0
  Supine diastolic BP increase from baseline >=20 mmHg | 1
  Supine diastolic BP decrease from baseline >=20 mmHg | 0
  Supine pulse rate value <40 bpm | 0
  Supine pulse rate value >120 bpm | 0
  Body temperature >38.5 °C | 0

17. Primary Outcome: Change From Baseline in Supine Systolic BP at Days 1, 2, 3, 4, 7, 14, 21 and 28
Description: BPs were assessed in a supine position with a completely automated device. Categorical classes for supine systolic BP of potential clinical concern included min value <90 mmHg, max decrease/increase from baseline >=30 mmHg.
Time Frame: Day 1 pre-dose (baseline); 1 hour, 2 hours, 4 hours, 8 hours and 12 hours post Day 1 dosing; Day 2; Day 3; Day 4; Day 7; Day 14; Day 21; Day 28.
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
mmHg
  1 hour post Day 1 dosing | 2.50 (9.503)
  2 hours post Day 1 dosing | 1.67 (8.189)
  4 hours post Day 1 dosing | 4.17 (8.519)
  8 hours post Day 1 dosing | -1.83 (5.981)
  12 hours post Day 1 dosing | 3.00 (9.274)
  Day 2 | -0.67 (6.346)
  Day 3 | 0.17 (8.183)
  Day 4 | 2.17 (4.446)
  Day 7 | 1.67 (10.053)
  Day 14 | 4.00 (7.563)
  Day 21 | 1.00 (8.854)
  Day 28 | -0.50 (13.019)

18. Primary Outcome: Change From Baseline in Diastolic Systolic BP at Days 1, 2, 3, 4, 7, 14, 21 and 28
Description: BPs were assessed in a supine position with a completely automated device. Categorical classes for supine diastolic BP of potential clinical concern included min value <50 mmHg, max decrease/increase from baseline >=20 mmHg.
Time Frame: as for outcome 17
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
mmHg
  1 hour post Day 1 dosing | -2.67 (7.659)
  2 hours post Day 1 dosing | -3.83 (7.910)
  4 hours post Day 1 dosing | -6.33 (7.146)
  8 hours post Day 1 dosing | -8.67 (6.653)
  12 hours post Day 1 dosing | -3.50 (8.597)
  Day 2 | -5.17 (6.145)
  Day 3 | -4.83 (8.085)
  Day 4 | -5.17 (6.145)
  Day 7 | -4.17 (9.087)
  Day 14 | 5.83 (9.475)
  Day 21 | -1.50 (8.118)
  Day 28 | -0.33 (6.218)

19. Primary Outcome: Change From Baseline in Supine Pulse Rate at Days 1, 2, 3, 4, 7, 14, 21 and 28
Description: Pulse rates were assessed in a supine position with a completely automated device. Categorical classes for supine pulse rate of potential clinical concern included min value <40 bpm or max value >120 bpm.
Time Frame: as for outcome 17
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
bpm
  1 hour post Day 1 dosing | -1.33 (3.011)
  2 hours post Day 1 dosing | -2.00 (3.521)
  4 hours post Day 1 dosing | 0.33 (11.003)
  8 hours post Day 1 dosing | -1.50 (11.537)
  12 hours post Day 1 dosing | -5.33 (6.501)
  Day 2 | -6.67 (8.937)
  Day 3 | -7.33 (6.683)
  Day 4 | -4.33 (11.361)
  Day 7 | 0.17 (15.198)
  Day 14 | 14.33 (12.209)
  Day 21 | 15.50 (13.882)
  Day 28 | 10.50 (12.740)

20. Primary Outcome: Change From Baseline in Oral Temperature at Days 1, 2, 3, 4, 7, 14, 21 and 28
Description: No eating, drinking, or smoking was allowed for 15 minutes prior to the measurement of oral temperature. The criterion for oral temperature of potential clinical concern was oral temperature > 38.5°C.
Time Frame: as for outcome 17
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
degree Celsius
  1 hour post Day 1 dosing | 0.10 (0.502)
  2 hours post Day 1 dosing | 0.28 (0.621)
  4 hours post Day 1 dosing | 0.50 (0.827)
  8 hours post Day 1 dosing | 0.17 (0.501)
  12 hours post Day 1 dosing | 0.22 (0.581)
  Day 2 | 0.25 (0.582)
  Day 3 | 0.10 (0.566)
  Day 4 | -0.08 (0.523)
  Day 7 | 0.30 (0.626)
  Day 14 | 0.45 (0.701)
  Day 21 | 0.67 (0.700)
  Day 28 | 0.75 (0.579)

21. Primary Outcome: Change From Baseline in Respiratory Rate at Days 1, 2, 3, 4, 7, 14, 21 and 28
Description: Respiratory rate measurement was preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Respiratory rate was measured in terms of "breaths per minute", and was measured by observing and counting the respirations of the participant for 30 seconds and multiplied by 2.
Time Frame: as for outcome 17
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
breaths per minute
  1 hour post Day 1 dosing | -0.50 (1.049)
  2 hours post Day 1 dosing | -0.67 (1.033)
  4 hours post Day 1 dosing | 0.17 (2.994)
  8 hours post Day 1 dosing | -0.50 (3.209)
  12 hours post Day 1 dosing | -1.50 (1.975)
  Day 2 | -1.33 (1.506)
  Day 3 | -1.67 (1.751)
  Day 4 | -1.67 (3.502)
  Day 7 | 1.00 (4.980)
  Day 14 | 3.50 (2.811)
  Day 21 | 3.83 (3.312)
  Day 28 | 2.67 (3.141)

22. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Categorical Criteria of Potential Clinical Concern
Description: Single 12-lead ECGs were performed for all participants in a supine position using an ECG machine that automatically calculated heart rate and measured PR, QRS and QT intervals. If a single time point ECG was abnormal, a triplicate ECG was required and obtained approximately 2-4 minutes apart; the average of triplicate ECG measurements collected at pre-dose Day 1 served as each participant's baseline value. Categorical classes for ECG data of potential clinical concern included: (1) QTcF - 450 millisecond (msec)≤ max value <480 msec, 480 msec ≤ max value <500 msec, max value ≥500 msec; 30 msec ≤ QTcF max increase from baseline <60 msec; max increase from baseline ≥60 msec; (2) PR interval - max value ≥300 msec, baseline value>200 and max increase from baseline ≥25%, baseline value ≤200 and max increase from baseline ≥50%; (3) QRS interval - max value ≥140 msec, increase from baseline ≥50%.
Time Frame: Day 1 to Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Participants
  PR Interval Value >=300 msec | 0
  PR Interval >=25% increase when baseline PR>200 msec, >=50% increase when baseline PR <=200 msec | 0
  QRS Interval value >=140 msec | 0
  QRS Interval % change from baseline >=50% | 0
  QT Interval value >500 msec | 0
  QTcF Interval value >= 450 msec and <480 msec | 0
  QTcF Interval value >= 480 msec and <500 msec | 0
  QTcF Interval value >= 500 msec | 0
  QTcF Interval change from baseline >=30 msec and <60 msec | 0
  QTcF Interval change from baseline >=60 msec | 0

23. Primary Outcome: Change From Baseline in ECG Mean Heart Rate at Days 1, 2, 3, 4, 7, 14, 21 and 28
Description: Heart rate was measured in terms of "beats per minute". Single 12-lead ECGs were performed for all participants in a supine position using an ECG machine that automatically calculated the heart rate and measured PR, QRS, and QT intervals. If a single time point ECG was abnormal, a triplicate ECG was required, which were obtained approximately 2-4 minutes apart; the average of the triplicate ECG measurements collected at pre-dose Day 1 served as each participant's baseline value.
Time Frame: as for outcome 17
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
beats per minute
  1 hour post Day 1 dosing | 0.43 (8.514)
  2 hours post Day 1 dosing | -1.57 (8.105)
  4 hours post Day 1 dosing | 1.43 (14.581)
  8 hours post Day 1 dosing | -1.73 (8.899)
  12 hours post Day 1 dosing | -1.57 (4.670)
  Day 2 | -3.07 (9.917)
  Day 3 | -3.90 (11.858)
  Day 4 | -5.73 (10.560)
  Day 7 | 0.60 (17.580)
  Day 14 | 9.43 (10.869)
  Day 21 | 3.60 (5.953)
  Day 28 | 4.43 (10.872)

24. Primary Outcome: Change From Baseline in PR Interval at Days 1, 2, 3, 4, 7, 14, 21 and 28
Description: Single 12-lead ECGs were performed for all participants in a supine position using an ECG machine that automatically calculated the heart rate and measured PR, QRS, and QT intervals. Categorical classes for PR interval data of potential clinical concern included: max value ≥300 ms, baseline value>200 and max increase from baseline≥25%, baseline value ≤200 and max increase from baseline ≥50%.
Time Frame: as for outcome 17
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
millisecond
  1 hour post Day 1 dosing | -4.22 (12.490)
  2 hours post Day 1 dosing | 0.45 (33.789)
  4 hours post Day 1 dosing | -8.38 (20.696)
  8 hours post Day 1 dosing | -6.55 (9.592)
  12 hours post Day 1 dosing | -10.88 (8.697)
  Day 2 | -2.72 (7.236)
  Day 3 | -6.05 (11.031)
  Day 4 | -4.55 (8.547)
  Day 7 | -6.22 (19.135)
  Day 14 | -10.22 (12.921)
  Day 21 | -8.05 (13.602)
  Day 28 | -4.05 (23.210)

25. Primary Outcome: Change From Baseline in QRS Interval at Days 1, 2, 3, 4, 7, 14, 21 and 28
Description: Single 12-lead ECGs were performed for all participants in a supine position using an ECG machine that automatically calculated the heart rate and measured PR, QRS, and QT intervals. Categorical classes for QRS interval data of potential clinical concern included: max value ≥140 ms, increase from baseline ≥50%.
Time Frame: as for outcome 17
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
millisecond
  1 hour post Day 1 dosing | -2.27 (4.698)
  2 hours post Day 1 dosing | -4.27 (6.953)
  4 hours post Day 1 dosing | -2.27 (5.972)
  8 hours post Day 1 dosing | -1.60 (4.459)
  12 hours post Day 1 dosing | 1.57 (5.315)
  Day 2 | -2.77 (7.640)
  Day 3 | -2.60 (5.713)
  Day 4 | -4.10 (5.968)
  Day 7 | -0.43 (4.855)
  Day 14 | -5.10 (5.312)
  Day 21 | -4.60 (5.646)
  Day 28 | -4.60 (7.505)

26. Primary Outcome: Change From Baseline in QT Interval at Days 1, 2, 3, 4, 7, 14, 21 and 28
Description: Single 12-lead ECGs were performed for all participants in a supine position using an ECG machine that automatically calculated the heart rate and measured PR, QRS, and QT intervals.
Time Frame: as for outcome 17
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
millisecond
  1 hour post Day 1 dosing | -6.57 (14.714)
  2 hours post Day 1 dosing | -0.90 (16.160)
  4 hours post Day 1 dosing | -11.07 (24.048)
  8 hours post Day 1 dosing | -0.07 (21.771)
  12 hours post Day 1 dosing | 2.60 (8.630)
  Day 2 | 0.77 (20.963)
  Day 3 | 0.60 (17.506)
  Day 4 | -0.07 (28.348)
  Day 7 | -5.90 (29.938)
  Day 14 | -30.40 (21.731)
  Day 21 | -17.57 (18.007)
  Day 28 | -19.07 (23.601)

27. Primary Outcome: Change From Baseline in QT Interval Corrected at Days 1, 2, 3, 4, 7, 14, 21 and 28
Description: Single 12-lead ECGs were performed for all participants in a supine position using an ECG machine that automatically calculated the heart rate and measured PR, QRS, and QT intervals. The corrected QT interval (QTc) estimates the QT interval at a standard heart rate of 60 bpm.
Time Frame: as for outcome 17
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
millisecond
  1 hour post Day 1 dosing | -4.15 (14.416)
  2 hours post Day 1 dosing | -4.82 (11.811)
  4 hours post Day 1 dosing | -7.15 (22.601)
  8 hours post Day 1 dosing | -4.15 (11.556)
  12 hours post Day 1 dosing | -0.32 (11.397)
  Day 2 | -7.82 (16.104)
  Day 3 | -11.65 (17.928)
  Day 4 | -16.82 (8.169)
  Day 7 | -4.98 (22.013)
  Day 14 | -8.48 (15.359)
  Day 21 | -8.98 (12.716)
  Day 28 | -8.65 (11.854)

28. Primary Outcome: Change From Baseline in Corrected QT Interval (Fridericia Method) (QTcF Interval) at Days 1, 2, 3, 4, 7, 14, 21 and 28
Description: Single 12-lead ECGs were performed for all participants in a supine position using an ECG machine that automatically calculated the heart rate and measured PR, QRS, and QT intervals. QTcF = QT interval corrected using the Fridericia method. Categorical classes for QTcF data of potential clinical concern included: 450 ms≤ max value <480 ms, 480≤ max value <500 ms, max value ≥500 ms; 30 ms ≤ QTcF max increase from baseline <60 ms; max increase from baseline ≥60 ms.
Time Frame: as for outcome 17
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
millisecond
  1 hour post Day 1 dosing | -5.38 (8.692)
  2 hours post Day 1 dosing | -3.22 (7.499)
  4 hours post Day 1 dosing | -8.55 (12.561)
  8 hours post Day 1 dosing | -2.88 (10.471)
  12 hours post Day 1 dosing | 0.28 (8.084)
  Day 2 | -4.88 (12.496)
  Day 3 | -7.05 (7.900)
  Day 4 | -10.88 (11.337)
  Day 7 | -5.55 (9.932)
  Day 14 | -15.22 (11.354)
  Day 21 | -11.05 (12.049)
  Day 28 | -11.38 (9.550)

29. Primary Outcome: Number of Participants With Physical Examination Findings
Description: A complete PE included assessments of the head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. A brief PE included assessments of the general appearance, the respiratory and cardiovascular systems, as well as participant reported symptoms. The full PE planned for Screening may have been performed on Day -1 before dosing at the discretion of the Investigator. If a full PE was done at Screening visit, a brief PE was to be conducted on Day-1. After Day -1, brief examinations based on signs and symptoms may have been performed if clinically indicated at the discretion of the Investigator to assess changes from baseline/previous visits of any ongoing symptoms.
Time Frame: Screening (Day -35 to Day -2), Day -1, Day 1 (for general appearance, heart, lungs), Day 7 (for general appearance, heart, lungs), Day 28 (for general appearance, heart, lungs)
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Participants
  Ears at screening | 0
  Ears on Day -1 | 0
  Eyes at screening | 0
  Eyes on Day -1 | 0
  Gastrointestinal at screening | 0
  Gastrointestinal on Day -1 | 0
  General appearance at screening | 0
  General appearance on Day -1 | 0
  General appearance on Day 1 | 0
  General appearance on Day 7 | 0
  General appearance on Day 28 | 0
  Head at screening | 0
  Head on Day -1 | 0
  Heart at screening | 0
  Heart on Day -1 | 0
  Heart on Day 1 | 0
  Heart on Day 7 | 0
  Heart on Day 28 | 0
  Lungs at screening | 0
  Lungs on Day -1 | 0
  Lungs on Day 1 | 0
  Lungs on Day 7 | 0
  Lungs on Day 28 | 0
  Lymph nodes at screening | 0
  Lymph nodes on Day -1 | 0
  Mouth at screening | 0
  Mouth on Day -1 | 0
  Musculoskeletal system at screening | 6
  Musculoskeletal system on Day -1 | 6
  Neurological system at screening | 0
  Neurological system on Day -1 | 0
  Nose at screening | 0
  Nose on Day -1 | 0
  Skin at screening | 0
  Skin on Day -1 | 0

30. Primary Outcome: Number of Participants With Injection Site Reactions
Description: Grades of injection site reactions were defined according to NCI CTCAE version 5.0. Grade 1=Tenderness with or without associated symptoms (eg, warmth, erythema, itching); Grade 2= Pain, lipodystrophy, edema, phlebitis; Grade 3= Ulceration or necrosis, severe tissue damage, operative intervention indicated; Grade 4=Life-threatening consequences, urgent intervention indicated; Grade 5=death. Participants with any grade of injection site reaction are reported in this outcome measure.
Time Frame: Day 1 to Day 7
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Participants | 0

31. Secondary Outcome: Mean Plasma Marstacimab Concentration Versus Time at Days 1, 2, 3, 4, 7, 14, 21 and 28
Description: Mean plasma concentration of marstacimab after participants received a single SC injection of marstacimab 300 mg.
Time Frame: Pre-dose, and 1 hour, 4 hours, 12 hours, 24 hours, 48 hours, 72 hours, and approximately 144 hours, 312 hours, 480 hours and 648 hours post Day 1 dosing
Population: The analysis population included all participants treated who had at least 1 marstacimab concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
ng/mL
  Day 1 pre-dose | 0.0000 (0.0000)
  1 hour post Day 1 dosing | 582.0 (1313.2)
  4 hours post Day 1 dosing | 1746 (960.3)
  12 hours post Day 1 dosing | 5647 (2254.2)
  Day 2, 24 hours post Day 1 dosing | 9033 (3349.8)
  Day 3, 48 hours post Day 1 dosing | 14300 (5510.3)
  Day 4, 72 hours post Day 1 dosing | 16060 (5706.9)
  Day 7, approximately 144 hours post Day 1 dosing | 14600 (4693.9)
  Day 14, approximately 312 hours post Day 1 dosing | 3437 (2349.3)
  Day 21, approximately 480 hours post Day 1 dosing | 53.17 (130.23)
  Day 28, approximately 648 hours post Day 1 dosing | 0.0000 (0.0000)

32. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Marstacimab
Description: Maximum plasma concentration of marstacimab after participants received a single SC injection of marstacimab 300 mg.
Time Frame: as for outcome 31
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention and had at least 1 of the PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
ng/mL | 15610 (35)

33. Secondary Outcome: Time for Cmax (Tmax) of Marstacimab
Description: Time for Cmax of marstacimab after participants received a single SC injection of marstacimab 300 mg.
Time Frame: as for outcome 31
Population: as for outcome 32
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
hour | 73.15 [71.9 to 167]

34. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Marstacimab
Description: Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration of marstacimab after participants received a single SC injection of marstacimab 300 mg.
Time Frame: as for outcome 31
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram * hour/milliliter (ng*hr/mL)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
nanogram * hour/milliliter (ng*hr/mL) | 2917000 (60)

35. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinity (AUCinf) of Marstacimab
Description: Area under the concentration time curve from time zero to infinity of marstacimab after participants received a single SC injection of marstacimab 300 mg.
Time Frame: as for outcome 31
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention and had at least 1 of the PK parameters. Number of Participants Analyzed = number of participants contributing to the summary statistics for this outcome measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 4
ng*hr/mL | 4549000 (7)

36. Secondary Outcome: Terminal Half-Life (t1/2) of Marstacimab
Description: Terminal half life (t1/2) of marstacimab after participants received a single SC injection of marstacimab 300 mg. t1/2 is defined as the time for plasma concentration to decrease by one half.
Time Frame: as for outcome 31
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 4
hour | 90.48 (26.025)

37. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Marstacimab
Description: Apparent volume of distribution of marstacimab after participants received a single SC injection of marstacimab 300 mg. Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F was influenced by the fraction absorbed. Vz/F was calculated as dose/AUCinf. AUCinf = area under the concentration time curve from time zero to infinity.
Time Frame: as for outcome 31
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 4
Liter | 8.305 (29)

38. Secondary Outcome: Apparent Clearance (CL/F) of Marstacimab
Description: Apparent clearance (CL/F) of marstacimab after participants received a single SC injection of marstacimab 300 mg. Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/F was calculated as Dose/ (AUCinf*kel). AUCinf = area under the concentration time curve from time zero to infinity. kel = terminal phase rate constant calculated by a linear regression of the log linear concentration time curve.
Time Frame: as for outcome 31
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 4
Liter per hour | 0.06595 (7)

39. Secondary Outcome: Maximum Increase From Baseline for Tissue Factor Pathway Inhibitor (TFPI), Day 1 up to Day 28
Description: TFPI is a protease inhibitor, which acts as an antagonist of the extrinsic coagulation pathway via inhibition of tissue factor-activated coagulation factor VII (FVIIa) and activated factor X (FXa). Plasma total TFPI levels were measured to reflect target binding with marstacimab. TFPI in results represented total TFPI.
Time Frame: Day 1 to Day 28
Population: The analysis population included all participants treated who had at least 1 of the pharmacodynamic (PD) parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
ng/mL | 79.50 (36.374)

40. Secondary Outcome: Area Under the Curve (AUC) of Change From Baseline Values (Days 1-7, Days 1-14, Days 1-28) for TFPI
Description: A change from baseline-time profile was established based on changes from baseline in TFPI at specific time points. Area under the TFPI change from baseline-time profile from time zero (Day 1) to Day 7, from time zero to Day 14 and from time zero to Day 28 are presented in this outcome measure. TFPI represented total TFPI.
Time Frame: as for outcome 31
Population: The analysis population included all participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
ng*hr/mL
  AUC of change from baseline values Days 1-7 for TFPI | 5730.07 (2891.283)
  AUC of change from baseline values Days 1-14 for TFPI | 15425.73 (9469.364)
  AUC of change from baseline values Days 1-28 for TFPI | 15526.33 (14100.382)

41. Secondary Outcome: Maximum Increase From Baseline for Prothrombin Fragments 1+2 (PF 1+2), Day 1 up to Day 28
Description: PF1+2 is an in vivo endpoint reflective of coagulation pathway activation. Maximum increase from baseline for PF 1+2 was provided.
Time Frame: Day 1 to Day 28
Population: All participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: picomole per liter (pmol/L)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
picomole per liter (pmol/L) | 531.9 (126.91)

42. Secondary Outcome: AUC of Change From Baseline Values (Days 1-7, Days 1-14, Days 1-28) for PF 1+2
Description: A change from baseline-time profile was established based on changes from baseline in PF 1+2 at specific time points. Area under the PF 1+2 change from baseline-time profile from time zero (Day 1) to Day 7, from time zero to Day 14 and from time zero to Day 28 are presented in this outcome measure.
Time Frame: as for outcome 31
Population: All participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: picomole * hour/liter (pmol*hr/L)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
picomole * hour/liter (pmol*hr/L)
  AUC of change from baseline values Days 1-7 for PF 1+2 | 56871.2823 (17578.69955)
  AUC of change from baseline values Days 1-14 for PF 1+2 | 116439.2948 (38634.76646)
  AUC of change from baseline values Days 1-28 for PF 1+2 | 144733.7020 (49783.67150)

43. Secondary Outcome: Maximum Increase From Baseline for D-Dimer, Day 1 up to Day 28
Description: D-dimer is an in vivo endpoint reflective of coagulation pathway activation. Maximum increase from baseline for D-Dimer is provided.
Time Frame: Day 1 to Day 28
Population: All participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (µg/mL)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
microgram per milliliter (µg/mL) | 0.463 (0.2881)

44. Secondary Outcome: AUC of Change From Baseline Values (Days 1-7, Days 1-14, Days 1-28) for D-Dimer
Description: A change from baseline-time profile was established based on changes from baseline in D-dimer at specific time points. Area under the D-dimer change from baseline-time profile from time zero (Day 1) to Day 7, from time zero to Day 14 and from time zero to Day 28 are presented in this outcome measure.
Time Frame: as for outcome 31
Population: The analysis population included all participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: microgram * hour/milliliter (µg*hr/mL)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
microgram * hour/milliliter (µg*hr/mL)
  AUC of change from baseline values Days 1-7 for D-dimer | 46.245 (29.3806)
  AUC of change from baseline values Days 1-14 for D-dimer | 110.855 (71.0567)
  AUC of change from baseline values Days 1-28 for D-dimer | 176.463 (153.1565)

45. Secondary Outcome: Maximum Decrease From Baseline for Dilute Prothrombin Time (dPT), Day 1 up to Day 28
Description: The dilute prothrombin time (dPT) is an ex vivo endpoint reflective of coagulation pathway activation. Maximum decrease from baseline for dPT is provided.
Time Frame: Day 1 to Day 28
Population: All participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: second
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
second | -19.62 (13.079)

46. Secondary Outcome: AUC of Change From Baseline Values (Days 1-7, Days 1-14, Days 1-28) for dPT
Description: A change from baseline-time profile was established based on changes from baseline in dPT at specific time points. Area under the dPT change from baseline-time profile from time zero (Day 1) to Day 7, from time zero to Day 14 and from time zero to Day 28 are presented in this outcome measure.
Time Frame: as for outcome 31
Population: The analysis population included all participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: second * hour (sec*hr)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
second * hour (sec*hr)
  AUC of change from baseline values Days 1-7 for dPT | -1910.10 (1800.853)
  AUC of change from baseline values Days 1-14 for dPT | -4079.87 (4094.644)
  AUC of change from baseline values Days 1-28 for dPT | -6792.18 (7068.384)

47. Secondary Outcome: Maximum Decrease From Baseline for Thrombin Generation Assay (TGA) Lag Time, Day 1 up to Day 28
Description: TGA lag time is an ex vivo endpoint reflective of coagulation pathway activation. Maximum decrease from baseline for TGA Lag Time is provided.
Time Frame: Day 1 to Day 28
Population: All participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
minute | -0.92 (0.279)

48. Secondary Outcome: AUC of Change From Baseline Values (Days 1-7, Days 1-14, Days 1-28) for TGA Lag Time
Description: A change from baseline-time profile was established based on changes from baseline in TGA lag time at specific time points. Area under the TGA lag time change from baseline-time profile from time zero (Day 1) to Day 7, from time zero to Day 14 and from time zero to Day 28 are presented in this outcome measure.
Time Frame: as for outcome 31
Population: The analysis population included all participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: minute * hour (min*hr)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
minute * hour (min*hr)
  AUC of change from baseline values Days 1-7 for TGA lag time | -95.10 (37.787)
  AUC of change from baseline values Days 1-14 for TGA lag time | -188.08 (81.227)
  AUC of change from baseline values Days 1-28 for TGA lag time | -174.70 (234.641)

49. Secondary Outcome: Maximum Increase From Baseline for TGA Peak, Day 1 up to Day 28
Description: TGA peak is an ex vivo endpoint reflective of coagulation pathway activation. Maximum increase from baseline for TGA Peak is provided.
Time Frame: Day 1 to Day 28
Population: All participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: nanomole (nmol)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
nanomole (nmol) | 105.83 (13.124)

50. Secondary Outcome: AUC of Change From Baseline Values (Days 1-7, Days 1-14, Days 1-28) for TGA Peak
Description: A change from baseline-time profile was established based on changes from baseline in TGA peak at specific time points. Area under the TGA peak change from baseline-time profile from time zero (Day 1) to Day 7, from time zero to Day 14 and from time zero to Day 28 are presented in this outcome measure.
Time Frame: as for outcome 31
Population: The analysis population included all participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: nanomole * hour (nmol*hr)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
nanomole * hour (nmol*hr)
  AUC of change from baseline values Days 1-7 for TGA peak | 10584.58 (3169.434)
  AUC of change from baseline values Days 1-14 for TGA peak | 20276.98 (5557.219)
  AUC of change from baseline values Days 1-28 for TGA peak | 28016.08 (9062.199)

51. Secondary Outcome: Maximum Increase From Baseline for TGA Endogenous Thrombin Potential (EGTP), Day 1 up to Day 28
Description: TGA EGTP is an ex vivo endpoint reflective of coagulation pathway activation. Maximum increase from baseline for TGA Endogenous Thrombin Potential is provided.
Time Frame: Day 1 to Day 28
Population: All participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: nanomole * minute (nmol*min)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
nanomole * minute (nmol*min) | 1093.7 (332.76)

52. Secondary Outcome: AUC of Change From Baseline Values (Days 1-7, Days 1-14, Days 1-28) for TGA EGTP
Description: A change from baseline-time profile was established based on changes from baseline in TGA EGTP at specific time points. Area under the TGA EGTP change from baseline-time profile from time zero (Day 1) to Day 7, from time zero to Day 14 and from time zero to Day 28 are presented in this outcome measure.
Time Frame: as for outcome 31
Population: The analysis population included all participants treated who had at least 1 of the PD parameters.
Measure: Mean (Standard Deviation); unit: nanomole * minute * hour (nmol*min*hr)
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
nanomole * minute * hour (nmol*min*hr)
  AUC of change from baseline values Days 1-7 for TGA EGTP | 123700.0 (35312.50)
  AUC of change from baseline values Days 1-14 for TGA EGTP | 238797.8 (47387.58)
  AUC of change from baseline values Days 1-28 for TGA EGTP | 332461.2 (69573.95)

53. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Against Marstacimab
Description: Summary of ADA incidence by visit is presented. ADA positive was defined as titer >=1.54.
Time Frame: Day 1 pre-dose (-2 hours to -5 min prior to dosing); Day 14; Day 21; Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 6
Participants
  Day 1 | 0
  Day 14 | 0
  Day 21 | 1
  Day 28 | 1

54. Secondary Outcome: Number of Participants With Neutralizing Antibody (NAb) Against Marstacimab
Description: Summary of NAb incidence by visit is presented. NAb positive was defined as titer >=1.08. ADA-positive participants (defined as titer >=1.54) were analyzed for NAb.
Time Frame: Day 1 pre-dose (-2 hours to -5 min prior to dosing); Day 14; Day 21; Day 28
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention. Number of Participants Analyzed = the total number of participants who had ADA-positive results in this study. Number Analyzed = Number of participants who had ADA-positive results at the specific time.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
Number analyzed (Participants) | 2
Participants
  Day 1: number analyzed (Participants) | 0
  Day 1 | 0
  Day 14: number analyzed (Participants) | 0
  Day 14 | 0
  Day 21: number analyzed (Participants) | 1
  Day 21 | 0
  Day 28: number analyzed (Participants) | 1
  Day 28 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to Day 42
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06741086 (Marstacimab) 300 mg Subcutaneous (SC) Single Dose (N=6)
Upper respiratory tract infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT04878731/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT04878731/SAP_001.pdf